CLINICAL TRIAL: NCT02493634
Title: Post-market Clinical Follow-up Study With Magnetic Resonance Imaging Conditional Guide Wire
Acronym: MRWIREPMCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nano4Imaging GmbH (Industry)
Collaborators: CERES GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N4IPMCF2015
Record Dates: First submitted 2015-06-22; First posted 2015-07-09 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Congenital Heart Defect
Keywords: Magnetic Resonance spectroscopy; Aortic Arch
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pressure gradient measurement (Other): Diagnostic procedure to measure pressure gradient in series of patients. Focus is on safety and absence of adverse events
  Interventions: Procedure: pressure gradient measurement; Device: MRWire

INTERVENTIONS:
Procedure: pressure gradient measurement — A guidewire is used to introduce and position a pressure catheter under magnetic resonance guidance to conduct flow and pressure measurement in the aortic arch to evaluate vascular resistance.
  Other Names: MRWire
Device: MRWire

SUMMARY:
This is post-market clinical follow-up study on 25 consecutive patients in two centers to evaluate the safety and performance of magnetic resonance imaging conditional guide wire and the acceptability of identified risks in the clinical evaluation and to detect emerging risks on the basis of factorial evidence.The procedure will be done in patients with a clinical indication for cardiac magnetic resonance and conventional catheterisation.

DETAILED DESCRIPTION:
This is post-market clinical follow-up study on 25 consecutive patients in two centers to evaluate the safety of a guide wire conditional for use in magnetic resonance imaging and the acceptability of identified risks in the clinical evaluation and to detect emerging risks on the basis of factorial evidence.

The guidewire is used to access the patients central circulatory system and in particular for the introduction and exact placement of a pressure catheter to measure the pressure gradient over the aortic arch. The procedure will be done in patients with a clinical indication for cardiac magnetic resonance and conventional catheterisation.Patients need to have a body weight over 40 kg and the introduction of a 5 French catheter should be possible. The primary endpoint is the measurement of procedural success, defined as successful insertion, steerability and visibility in MRI, in the absence of device related adverse events such as damage to vessel wall. In addition structural integrity of the instruments is to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical indication for cardiac magnetic resonance and conventional diagnostic catheterisation
* patients with body weight of > 40 kg in which the introduction of an introducer of > 5 French is possible.
* subject provided written informed consent using the approved consent form or in case of a minor the subject provided written assent and its legal guardian provided written informed consent.

Exclusion Criteria:

* major surgery in the last 42 days
* history of irreversible bleeding disorder
* contraindication to cardiac magnetic resonance
* Contraindications to guidewire procedures, such as evidence of active infection
* women of child-bearing potential who cannot provide a negative pregnancy test
* chronic total occlusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-18 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Procedural success | Up to 30 days after procedure
  procedural success means that insertion, steerability and visibility of the guide wire in the MR guided intervention was successfully reached, in the absence of adverse events up to 30 days after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ewert, Prof, MD, Principal Investigator — German Heart Center
Locations (3):
- Germany (2):
  - Deutsches Herzzentrum Munchen, Munich, Bavaria
  - Herzzentrum Leipzig, Leipzig
- Royal Free Hospital- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kos S, Huegli R, Hofmann E, Quick HH, Kuehl H, Aker S, Kaiser GM, Borm PJ, Jacob AL, Bilecen D. First magnetic resonance imaging-guided aortic stenting and cava filter placement using a polyetheretherketone-based magnetic resonance imaging-compatible guidewire in swine: proof of concept. Cardiovasc Intervent Radiol. 2009 May;32(3):514-21. doi: 10.1007/s00270-008-9483-5. Epub 2008 Dec 30. PMID 19115070
- [Background] Kos S, Huegli R, Hofmann E, Quick HH, Kuehl H, Aker S, Kaiser GM, Borm PJ, Jacob AL, Bilecen D. MR-compatible polyetheretherketone-based guide wire assisting MR-guided stenting of iliac and supraaortic arteries in swine: feasibility study. Minim Invasive Ther Allied Technol. 2009;18(3):181-8. doi: 10.1080/13645700902921971. PMID 19431070
- [Background] Kos S, Huegli R, Hofmann E, Quick HH, Kuehl H, Aker S, Kaiser GM, Borm PJ, Jacob AL, Bilecen D. Feasibility of real-time magnetic resonance-guided angioplasty and stenting of renal arteries in vitro and in Swine, using a new polyetheretherketone-based magnetic resonance-compatible guidewire. Invest Radiol. 2009 Apr;44(4):234-41. doi: 10.1097/RLI.0b013e31819b00f1. PMID 19252440